CLINICAL TRIAL: NCT00415428
Title: Patient And Physician Alliance -Guideline Education Treatment Optimization
Brief Title: A Quality Ensuring Project With Focus On Patients With Cardiovascular Diseases As Well As Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581154
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Heart Diseases; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1.
  Interventions: Behavioral: Patient adherence to national educational guidelines.

INTERVENTIONS:
Behavioral: Patient adherence to national educational guidelines.

SUMMARY:
The overall objective is to increase the adherence to national guidelines for patients with established CVD and/or Type 2 diabetes by means of repeated post-graduate educational meetings and regular evaluation of the optimisation initiatives, demonstrated by improvement of goal attainment in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to meet all of the inclusion criteria to be eligible for enrollment into the study. The following subjects qualify for inclusion in the study:
* Subjects for whom measurement of total cholesterol, low density lipoprotein (LDL) cholesterol, blood pressure (BP) and glycosylated hemoglobin (HbA1c) was planned independently of this observational study and for whom baseline values were or became available.
* Subjects with known CVD diagnosed > or = 6 months before inclusion
* Previous myocardial infarction
* Ischemic heart disease (stable and unstable angina pectoris)
* Ischemic apoplexy
* Peripheral arterial disease
* And/Or
* Subjects with T2D diagnosed > or = 6 months before inclusion
* At least 50% of the subjects had to have CVD as the primary diagnosis. It was allowed for a secondary diagnosis to be <6 months before inclusion.

Exclusion Criteria:

* Subjects presenting with any of the following were not to be included in the study:
* Life expectancy of < or = 2 years
* Unable/unwilling to understand/follow instructions
* Taking part in a clinical study involving an investigational drug
* Followed by a specialist for their CVD and/or T2D at the time of inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic patients
Sampling Method: Probability Sample
Enrollment: 2776 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581154&StudyName=A%20Quality%20Ensuring%20Project%20With%20Focus%20On%20Patients%20With%20Cardiovascular%20Diseases%20As%20Well%20As%20Type%202%20Diabetes.